CLINICAL TRIAL: NCT01133626
Title: A Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel-Group, 6-Week Study Designed to Investigate the Effects of BDP HFA Nasal Aerosol on the Hypothalamic-Pituitary-Adrenal (HPA) Axis When Administered in Adolescent and Adult Subjects (12 to 45 Years of Age) With Perennial Allergic Rhinitis (PAR)
Brief Title: Hypothalamic-Pituitary-Adrenal (HPA) Axis Study in Adult and Adolescent Subjects With Perennial Allergic Rhinitis (PAR)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BDP-AR-304
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-05

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Prednisone; Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants self-administered 4 actuations (two per nostril) of placebo HFA once daily each morning for 6 weeks (42 days) as double-blind therapy for BDP. During week 6 (days 36-42), participants also took a placebo capsule as double-blind therapy for prednisone.
  Interventions: Drug: Placebo Nasal Aerosol; Drug: Placebo Prednisone Capsules
- BDP HFA 320 µg/day (Experimental): Participants self-administered 4 actuations (two per nostril) of 80 µg BDP HFA once daily each morning for 6 weeks (42 days). During week 6 (days 36-42), participants also took a placebo capsule as double-blind therapy for prednisone.
  Interventions: Drug: Placebo Prednisone Capsules; Drug: Beclomethasone dipropionate
- Prednisone (Active Comparator): Participants self-administered 4 actuations (two per nostril) of placebo HFA once daily each morning for 6 weeks (42 days) as double-blind therapy for BDP. During week 6 (days 36-42), participants also took a 10/mg a day prednisone capsule.
  Interventions: Drug: Placebo Nasal Aerosol; Drug: Prednisone capsules

INTERVENTIONS:
Drug: Placebo Nasal Aerosol — Placebo nasal aerosol administered daily for 42 days of treatment
  Arms: Placebo; Prednisone
Drug: Prednisone capsules — Prednisone 10 mg capsule taken each day on the last 7 days of treatment
  Arms: Prednisone
Drug: Placebo Prednisone Capsules — Placebo prednisone capsule taken each day on the last 7 days of treatment
  Arms: BDP HFA 320 µg/day; Placebo
Drug: Beclomethasone dipropionate — Total daily dose of 320 micrograms per day of beclomethasone dipropionate (BDP) hydrofluoroalkane (HFA) applied as a nasal aerosol each morning for 42 days.
  Other Names: QNASL(TM)
  Arms: BDP HFA 320 µg/day

SUMMARY:
The purpose of the study is to evaluate the effects of BDP HFA Nasal Aerosol on HPA-axis function.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Male or female subjects 12-45 years of age
* Documented history of perennial allergic rhinitis
* General good health
* Other criteria apply

Exclusion Criteria:

* History of physical findings of nasal pathology (within 60 days prior to Screening Visit 1)
* Participation in any investigational drug study 30 days preceding Screening Visit 1
* History of respiratory infection/disorder with 14 days preceding Screening Visit 1
* Use of any prohibited concomitant medications

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudeesh K. Tantry, Ph.D., Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (3):
- United States (3):
  - Teva Clinical Study Site, North Dartmouth, Massachusetts
  - Teva Clinical Study Site, New Braunfels, Texas
  - Teva Clinical Study Site, San Antonio, Texas

REFERENCES:
- [Result] Hampel FC, Ratner PH, Miller SD, Melchior A, Dunbar SA, Tantry SK, Dorinsky PM. Once-daily treatment with beclomethasone dipropionate hydrofluoroalkane nasal aerosol (320 mcg/d) is not associated with hypothalamic-pituitary-adrenal axis suppression in adolescent subjects with perennial allergic rhinitis. J Allergy Clin Immunol 2012; 129:AB188
- [Result] Ratner PH, Miller SD, Hampel FC, A, Dunbar SA, Tantry SK, Dorinsky PM (2011). BDP HFA Nasal Aerosol 320 μg Once Daily g Once Daily Is Not Associated with HPA-Axis Suppression in Subjects With Perennial Allergic Rhinitis. Ann Allergy Asthma Immunol. 107(11):A118.
- [Derived] Ratner PH, Miller SD, Hampel FC Jr, Melchior A, Dunbar SA, Tantry SK. Once-daily treatment with beclomethasone dipropionate nasal aerosol does not affect hypothalamic-pituitary-adrenal axis function. Ann Allergy Asthma Immunol. 2012 Nov;109(5):336-41. doi: 10.1016/j.anai.2012.08.005. PMID 23062389

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 139 patients were screened and 128 patients were enrolled in the study and participated in the Run-in Period. Of the 128 enrolled patients, 107 were randomized to study treatment.
Pre-assignment Details: During the 7 to 14 day Run-in Period (prior to randomization), participants self-administered a single-blind placebo nasal aerosol once daily in the morning.
Groups:
- BDP HFA 320 µg/Day: Participants self-administered 4 actuations (two per nostril) of 80 µg beclomethasone dipropionate (BDP) hydrofluoroalkane (HFA) once daily each morning for 6 weeks (42 days). During week 6 (days 36-42), participants also took a placebo capsule as double-blind therapy for prednisone.
- Placebo/Prednisone: Participants self-administered 4 actuations (two per nostril) of placebo HFA once daily each morning for 6 weeks (42 days) as double-blind therapy for BDP. During week 6 (days 36-42), participants also took a 10/mg a day prednisone capsule.
Period: Overall Study
Arm/Group | BDP HFA 320 µg/Day | Placebo | Placebo/Prednisone
Started | 50 | 46 | 11
Safety Population | 50 (Participants who received at least 1 dose of study drug) | 46 (Participants who received at least 1 dose of study drug) | 11 (Participants who received at least 1 dose of study drug)
Per Protocol Population | 48 (Received >=1 dose of study drug and >=1 post-baseline assessment prior to major protocol deviation.) | 41 (Received >=1 dose of study drug and >=1 post-baseline assessment prior to major protocol deviation.) | 9 (Received >=1 dose of study drug and >=1 post-baseline assessment prior to major protocol deviation.)
Completed | 49 | 41 | 9
Not Completed | 1 | 5 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Other | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BDP HFA 320 µg/Day | Placebo | Placebo/Prednisone | Total
Number analyzed (Participants) | 48 | 41 | 9 | 98
Age Continuous [Mean (Standard Deviation); unit: years] — Demographic data are provided for the Per Protocol population.
  years | 28.3 (10.0) | 26.6 (10.6) | 26.2 (11.9) | 27.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 7 | 54
  Male | 23 | 19 | 2 | 44
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 18 | 17 | 2 | 37
  Not Hispanic or Latino | 30 | 24 | 7 | 61
Race/Ethnicity, Customized [Number; unit: participants] — A participant may select more than one race type.
  participants
    American Indian or Alaska Native | 0 | 0 | 1 | 1
    Asian | 1 | 0 | 0 | 1
    Black or African American | 7 | 2 | 1 | 10
    White | 42 | 38 | 7 | 87
    Unknown or Not Reported | 0 | 1 | 0 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (7.9) | 27.0 (6.2) | 28.4 (7.9) | 27.6 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: The 24-hour Serum Cortisol Weighted Mean After 42 Days of Treatment
Description: Geometric mean serum cortisol weighted mean values were calculated at baseline and after 6 weeks (42 days) of treatment. The geometric mean ratio of week 6 / baseline is reported. The primary outcome compares the BDP HFA and Placebo treatment arms. The comparison of active control (Placebo/Prednisone) and Placebo treatment arms is an "other pre-specified" outcome.
Time Frame: Day 0 (Baseline), Day 42
Population: Per protocol population
Measure: Geometric Mean (Standard Error); unit: ratio
Arm/Group | BDP HFA 320 µg/Day | Placebo | Placebo/Prednisone
Number analyzed (Participants) | 48 | 41 | 9
ratio | 0.90 (1.04) | 0.95 (1.03) | 0.31 (1.14)
Statistical Analysis 1: Comparison: BDP HFA 320 µg/Day vs Placebo; Test type: Non-Inferiority or Equivalence — Non-inferiority would be demonstrated if the lower limit of a two-sided 95% CI for the geometric mean ratio of BDP HFA 320 mcg/day to placebo was greater than 0.80; ANCOVA; geometric mean ratio = 0.96, 95% CI 2-sided [0.87 to 1.06]

ADVERSE EVENTS:
Arm/Group | BDP HFA 320 µg/Day | Placebo | Placebo/Prednisone
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/46 | 0/11
Other Adverse Events (participants affected / at risk) | 3/50 | 3/46 | 5/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BDP HFA 320 µg/Day (N=50) | Placebo (N=46) | Placebo/Prednisone (N=11)
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Blood oestrogen increased (Investigations) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.